CLINICAL TRIAL: NCT00752206
Title: A Randomized, Double-Blinded, Placebo-Controlled, Multi-Institutional, Cross-over, Phase II.5 Study of Saracatinib (AZD0530), a Selective Src Kinase Inhibitor, In Patients With Recurrent Osteosarcoma Localized to the Lung
Brief Title: A Placebo-Controlled Study of Saracatinib (AZD0530) in Patients With Recurrent Osteosarcoma Localized to the Lung
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Data Safety Monitoring Board (DSMB) recommended study termination for slow accrual and futility.
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SARC012; D8180C00039; NCT00923286 (obsolete NCT alias)
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-04

CONDITIONS: Osteosarcoma
Keywords: AZD0530; Saracatinib; Osteosarcoma; Recurrent; Localized; to the Lung
MeSH Terms: conditions — Osteosarcoma; Recurrence | interventions — saracatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saracatinib (Active Comparator): Saracatinib will be administered as a once daily, oral dose of 175 mg, for a 28-day cycle, with no breaks between cycles. The duration of treatment with saracatinib will be 13 cycles.
  Interventions: Drug: Saracatinib
- Placebo (Placebo Comparator): Placebo will be administered as a once daily, oral dose of 175 mg, for a 28-day cycle, with no breaks between cycles. The duration of treatment with placebo will be 13 cycles.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saracatinib — Oral Agent
  Arms: Saracatinib
Drug: Placebo — Oral Agent
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine how long patients who undergo complete surgical removal of recurrent osteosarcoma in the lung will remain free of cancer after taking Saracatinib compared to patients taking placebo (a sugar pill).

DETAILED DESCRIPTION:
Further details provided by SARC (Sarcoma Alliance for Research through Collaboration):

After complete surgical removal of their cancer, patients will be randomly assigned to receive either Saracatinib or placebo (a sugar pill) throughout the study. Patients will take Saracatinib (or placebo) once daily by mouth for a total of 364 days. The duration of treatment is divided into 13 cycles, 28 days each cycle with no breaks in between.

Patients will be seen for interim medical history, physical exam and laboratory studies prior to each cycle. To monitor for recurrence of tumor, patients will undergo thoracic CT scans at 3-4 weeks, 6-8 weeks, at 3 months, at 6 months, at 9 months, at 12 months, then every 6 months up to 2 years, and then every year up to 5 years after starting treatment. An electrocardiogram (ECG) will be taken at 3 months, and a bone scan will be performed at 12 months.

Patients who recur in the lung while on-study and who are thought to be amenable to complete surgical resection will be able to find out if they were receiving placebo or saracatinib. Those patients who were receiving placebo may then have the option of undergoing surgical resection. If fully resected of all recurrent disease,they will be given the option of receiving oral therapy with saracatinib. Saracatinib will be administered as a once daily, oral dose of 175 mg, for a 28-day cycle, with no breaks between cycles. The duration of treatment with saracatinib will be thirteen 28-day cycles (364 days total). If complete resection of all lung nodules is not achieved, the patient will be removed from the study.

Patients who recur in locations other than the lung while on-study will be taken off study at that time.

Blood and tumor samples for research purposes will be collected at the time the tumor is removed.

After completing all 13 cycles, patients will be followed for approximately every 3 months until 2 years from starting treatment, then approximately every 6 months until 4 years from starting treatment, and once at year 5.

ELIGIBILITY:
Inclusion Criteria:

* Patient had recurrence of osteosarcoma, localized to the lungs, had complete surgical removal of all lung nodules are eligible for enrollment.
* Patient with suspected recurrence of osteosarcoma but who has not had surgery is eligible for enrollment but will not be randomized to receive study medication until deemed fully eligible following surgical removal of all lung nodules.
* Patient had histological confirmed diagnosis of osteosarcoma of the recurrent sample.
* Patient had recurrence of osteosarcoma in the lung following standard therapy including: adriamycin, cisplatin, ifosfamide and methotrexate.
* Patient is ≥ 15 and < 75 years of age.
* Weight ≥ 34 kg.
* ECOG performance score of 0-2.
* Adequate bone marrow function.
* Adequate renal function.
* Adequate hepatic function.
* Adequate cardiac function.
* Women of childbearing potential must have had a negative pregnancy test (urine or serum) ≤ 7 days prior to enrollment, and willingness to use an acceptable method of contraception during participation in the study and for 3 months after the last dose.
* Randomization must occur ≤ 6 weeks after complete surgical resection.
* Patient or legal guardian has signed informed consent.

Exclusion Criteria:

* Presence of metastatic disease in other locations in addition to the lung.
* Disruption of the lung pleura by tumor.
* Paget's disease.
* Patient currently using, or has previously used CYP3A4 inducers or inhibitors within 2 to 14 days prior to the initiation of oral therapy.
* Known hypersensitivity to other Src/Abl non-receptor kinase inhibitors.
* Evidence of interstitial lung disease.
* Any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol.
* Myocardial infarction within one year prior to study entry.
* Bleeding diathesis, resulting in symptomatic bleeding.
* Patient is pregnant or nursing/breast-feeding.
* Patient received chemotherapy, biological or investigational agent ≤ 28 days prior to enrollment.
* Patient experiencing unresolved toxicity ≥ CTCAE grade 2 (except alopecia) from previous agents.

Ages: 15 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Baird, MD, Principal Investigator — National Cancer Institute - Pediatric Oncology Branch
Locations (18):
- United States (18):
  - University of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - UCLA/Mattel's Children's Hospital, Los Angeles, California
  - Stanford University, Palo Alto, California
  - UCSF, San Francisco, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - National Cancer Institute, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Cancer Care Alliance/University of Washington Medical Center, Seattle, Washington

REFERENCES:
- See also: Related Info — http://www.sarctrials.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Saracatinib: Saracatinib: Oral Agent
  Administered once daily, oral dose of 175 mg for a 28 day cycle.
- Placebo: Placebo
  Administered once daily, oral dose of 175 mg for a 28 day cycle.
Period: Overall Study
Arm/Group | Saracatinib | Placebo
Started | 19 | 19
Completed | 10 | 8
Not Completed | 9 | 11
Not completed — Disease progression | 8 | 11
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Population: 38 subjects were randomized to receive therapy. One subject was taken off study for pregnancy, therefore 37 subjects were included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saracatinib | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 23.89 (8.53) | 26.63 (12.07) | 25.30 (10.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 11 | 8 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 12 | 14 | 26
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 14 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 8
Histology types [Count of Participants; unit: Participants] — Population: 38 subjects were randomized to receive therapy. One subject was taken off study for pregnancy, therefore 37 subjects were included in the analysis.
  Participants
    Osteoblastic sub-type | 9 | 12 | 21
    Chondroblastic | 6 | 3 | 9
    Telangiectatic | 3 | 1 | 4
    Fibroblastic | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate Among Patients Treated With Saracatinib and Placebo.
Description: To determine if the addition of saracatinib to pulmonary metastasectomy, versus placebo and pulmonary metastasectomy, results in a change in progression free survival.
Time Frame: Evaluation for recurrence/progression will be made every 3 months for the 1st year, then every 6 months up to 2 years, then every year up to 5 years after starting treatment.
Population: 38 subjects were randomized to receive therapy. One randomized subject was subsequently taken off-study for pregnancy; therefore 37 subjects were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Saracatinib | Placebo
Number analyzed (Participants) | 18 | 19
months | 19.4 [0 to 60] | 8.6 [0 to 60]

2. Secondary Outcome: Change in Overall Survival With the Addition of Saracatinib to Pulmonary Metastasectomy, Versus Placebo and Pulmonary Metastasectomy
Description: To determine if the addition of saracatinib to pulmonary metastasectomy, versus placebo and pulmonary metastasectomy, results in a change in overall survival.
Time Frame: 5 year overall survival
Measure: Median (85% Confidence Interval); unit: months
Arm/Group | Saracatinib | Placebo
Number analyzed (Participants) | 18 | 19
months | NA [45 to 70] — Median overall survival (OS) not reached in either group and the curves overlapped. | NA [45 to 70] — Median overall survival (OS) not reached in either group and the curves overlapped.

3. Secondary Outcome: Change in Time to Treatment Failure With the Addition of Saracatinib to Pulmonary Metastasectomy, Versus Placebo and Pulmonary Metastasectomy
Description: To determine if the addition of saracatinib to pulmonary metastasectomy, versus placebo and pulmonary metastasectomy, results in a change in the time to treatment failure. Time to treatment failure is the time from randomization to treatment discontinuation.
Time Frame: Up to 12 months
Population: Did not perform time to progression analysis, but rather evaluated PFS. There was no data to report for time to treatment failure.
Arm/Group | Saracatinib | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Genes Identified for Prediction of Recurrence of Osteosarcoma
Description: To perform microarray analysis of tumor samples to identify a gene signature that predicts for recurrence of osteosarcoma using methodology that relies on preparation of RNA, followed by cDNA. Fluorescent labeling followed by hybridization to a DNA chip allows for quantitative scanning for hybridized complexes.
Time Frame: Up to 12 months
Measure: Number; unit: identified genes
Arm/Group | Saracatinib | Placebo
Number analyzed (Participants) | 18 | 19
identified genes | 0 | 0

5. Secondary Outcome: Biomarkers Related to Activation of Src and Src Substrates
Description: To evaluate tumor samples for biomarkers related to activation of Src and Src substrates.
Time Frame: Up to 12 months
Population: This testing was not performed.
Arm/Group | Saracatinib | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Cell Lines and Murine Xenografts From Recurrent Tumor Samples
Description: To establish cell lines and murine xenografts from recurrent tumor samples.
Time Frame: Up to 12 months
Population: This testing was not performed.
Arm/Group | Saracatinib | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Mutations Identified That May be Causative For Recurrent Osteosarcoma
Description: To perform sequencing analysis of DNA and RNA in tumor samples compared to normal blood to detect mutations that may be causative for recurrent osteosarcoma. The methodology uses transcriptome sequencing, exon re-sequencing and mate-pair end sequencing, allowing us to detect translocations. The availability of matched normal DNA in the blood will allow us to determine which changes are unique to the tumor.
Time Frame: Up to 12 months
Measure: Number; unit: identified mutations
Arm/Group | Saracatinib | Placebo
Number analyzed (Participants) | 18 | 19
identified mutations | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 years
Groups:
- Placebo: Administered once daily, oral dose of 175 mg for a 28 day cycle.
Arm/Group | Saracatinib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/18 | 2/19
Other Adverse Events (participants affected / at risk) | 18/37 | 19/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saracatinib (N=18) | Placebo (N=19)
Lung Nodules (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Glioblastoma Multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Saracatinib (N=37) | Placebo (N=37)
Abdominal pain (Gastrointestinal disorders) | 3/18 | 2/19
Acne (Skin and subcutaneous tissue disorders) | 2/18 | 1/19
Alanine Aminotransferase increased (Investigations) | 3/18 | 3/19
Alkaline Phosphatase increased (Investigations) | 4/18 | 3/19
Allergic reaction (Immune system disorders) | 1/18 | 0/19
Alopecia (Skin and subcutaneous tissue disorders) | 1/18 | 0/19
Amylase increased (Investigations) | 1/18 | 0/19
Anorexia (Metabolism and nutrition disorders) | 1/18 | 2/19
Arthritis (Musculoskeletal and connective tissue disorders) | 0/18 | 1/19
Aspartate aminotransferase increased (Investigations) | 5/18 | 2/19
Asthma (Respiratory, thoracic and mediastinal disorders) | 1/18 | 0/19
Back pain (Musculoskeletal and connective tissue disorders) | 2/18 | 1/19
Breast pain (Reproductive system and breast disorders) | 0/18 | 1/19
Bruising (Injury, poisoning and procedural complications) | 1/18 | 0/19
Chest pain (General disorders) | 1/18 | 0/19
Flu like symptoms (General disorders) | 1/18 | 0/19
Cough (Respiratory, thoracic and mediastinal disorders) | 3/18 | 4/19
CPK increased (Investigations) | 1/18 | 0/19
Creatinine increased (Investigations) | 2/18 | 2/19
Depression (Psychiatric disorders) | 1/18 | 0/19
Dermatology/Skin- Other (Skin and subcutaneous tissue disorders) | 2/18 | 0/19
Diarrhea (Gastrointestinal disorders) | 6/18 | 4/19
Dizziness (Nervous system disorders) | 2/18 | 0/19
Dry skin (Skin and subcutaneous tissue disorders) | 2/18 | 0/19
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/18 | 0/19
Hyperparathyroidism (Endocrine disorders) | 1/18 | 0/19
Gastroenteritis (Respiratory, thoracic and mediastinal disorders) | 1/18 | 1/19
External ear pain (Ear and labyrinth disorders) | 0/18 | 1/19
Eye pain (Eye disorders) | 1/18 | 0/19
Fatigue (General disorders) | 4/18 | 5/19
Fever (General disorders) | 2/18 | 1/19
Flushing (Vascular disorders) | 1/18 | 0/19
Fracture (Injury, poisoning and procedural complications) | 0/18 | 1/19
Gastrointestinal- Other (Gastrointestinal disorders) | 0/18 | 1/19
Gingival pain (Gastrointestinal disorders) | 0/18 | 1/19
Headache (Nervous system disorders) | 3/18 | 5/19
Hearing impaired (Ear and labyrinth disorders) | 1/18 | 0/19
Heartburn (Gastrointestinal disorders) | 2/18 | 0/19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2/18 | 1/19
Hot flashes (Vascular disorders) | 0/18 | 1/19
Hyperbilirubinemia (Investigations) | 1/18 | 1/19
Hyperglycemia (Metabolism and nutrition disorders) | 5/18 | 4/19
Hypermagnesemia (Metabolism and nutrition disorders) | 3/18 | 1/19
Hypertension (Vascular disorders) | 0/18 | 1/19
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1/18 | 0/19
Hypoalbuminemia (Metabolism and nutrition disorders) | 1/18 | 0/19
Hypocalcemia (Metabolism and nutrition disorders) | 2/18 | 0/19
Hypoglycemia (Metabolism and nutrition disorders) | 2/18 | 2/19
Hypokalemia (Metabolism and nutrition disorders) | 1/18 | 2/19
Hypomagnesemia (Metabolism and nutrition disorders) | 1/18 | 2/19
Hyponatremia (Metabolism and nutrition disorders) | 0/18 | 2/19
Hypophosphatemia (Metabolism and nutrition disorders) | 7/18 | 7/19
Upper respiratory infection (Infections and infestations) | 3/18 | 3/19
Insomnia (Psychiatric disorders) | 1/18 | 1/19
Constipation (Gastrointestinal disorders) | 0/18 | 1/19
Joint pain (Musculoskeletal and connective tissue disorders) | 2/18 | 1/19
Groin pain (Musculoskeletal and connective tissue disorders) | 1/18 | 0/19
Leukopenia (Investigations) | 5/18 | 2/19
Lymphopenia (Investigations) | 2/18 | 2/19
Mucositis (Gastrointestinal disorders) | 0/18 | 2/19
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2/18 | 0/19
Myalgia (Musculoskeletal and connective tissue disorders) | 1/18 | 2/19
Nail thinning (Skin and subcutaneous tissue disorders) | 1/18 | 0/19
Nausea (Gastrointestinal disorders) | 6/18 | 3/19
Neutropenia (Investigations) | 3/18 | 0/19
Ocular-Other (Eye disorders) | 0/18 | 1/19
Oculomotor nerve disorder (Nervous system disorders) | 1/18 | 0/19
Middle ear infection (Infections and infestations) | 1/18 | 1/19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/18 | 4/19
Muscle pain (Musculoskeletal and connective tissue disorders) | 1/18 | 0/19
Neck pain (Musculoskeletal and connective tissue disorders) | 1/18 | 0/19
Back pain (Musculoskeletal and connective tissue disorders) | 1/18 | 1/19
Stomach pain (Gastrointestinal disorders) | 1/18 | 0/19
Palpitations (Cardiac disorders) | 0/18 | 1/19
Peripheral sensory neuropathy (Nervous system disorders) | 1/18 | 1/19
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2/18 | 2/19
Thrombocytopenia (Investigations) | 4/18 | 3/19
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1/18 | 0/19
Concentration impairment (Nervous system disorders) | 0/18 | 1/19
Proteinuria (Renal and urinary disorders) | 0/18 | 1/19
Pruritus (Skin and subcutaneous tissue disorders) | 1/18 | 0/19
Activated partial thromboplastin time prolonged (Investigations) | 0/18 | 1/19
Pulmonary- Other (Respiratory, thoracic and mediastinal disorders) | 0/18 | 1/19
Rash (Skin and subcutaneous tissue disorders) | 4/18 | 3/19
Rectal hemorrhage (Gastrointestinal disorders) | 1/18 | 0/19
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 3/18 | 2/19
Rigors/chills (General disorders) | 1/18 | 0/19
Ulceration in right nare (Respiratory, thoracic and mediastinal disorders) | 1/18 | 0/19
Vitamin D deficiency (Investigations) | 0/18 | 1/19
Vomiting (Gastrointestinal disorders) | 2/18 | 1/19
Weight loss (Investigations) | 1/18 | 0/19
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 1/18 | 0/19
Anemia (Blood and lymphatic system disorders) | 3/18 | 2/19
Sexual-Other (Reproductive system and breast disorders) | 0/18 | 1/19
Small groundglass focus of airspace disease (Respiratory, thoracic and mediastinal disorders) | 0/18 | 1/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-09-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT00752206/Prot_SAP_000.pdf